CLINICAL TRIAL: NCT03804437
Title: The Prevalence and Anatomical Variations of Bifid Mandibular Canal in a Sample of Egyptian Population Using CBCT.A Hospital-based Cross-Sectional Study
Brief Title: The Prevalence and Anatomical Variations of Bifid Mandibular Canal in the Egyptian Population Using Cone Beam CT (CBCT)
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Enas El Saket, Master degree student, Cairo University
Other Study IDs: ORAD 7-1-1
Record Dates: First submitted 2019-01-07; First posted 2019-01-15 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: The Prevalence of Bifid Mandibular Canal
Keywords: Mandibular canals; bifid canal; cbct; cbct dental.

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The prevalence of bifid mandibular canal will be detected in a sample of Egyptian Population.Anatomical variations of the bifid canal will also be detected.

DETAILED DESCRIPTION:
Settings:

The data collection will be obtained from the data base available at the department of Oral and Maxillofacial Radiology, Faculty of Dentistry, Cairo University. CBCT images will be obtained from Egyptian patients who were referred to the CBCT unit in oral and maxillofacial radiology department for different purposes.

Variables:

•Prevalence of bifid canals - Classification and prevalence of observed types - Distance from the involved teeth

Data Sources / Measurements:

* Retrospective Data Analysis will be performed after the CBCT images are pooled from the computer database.
* Exposure parameters of the scans will vary depending on patients' sizes (according to the manufacturer's recommendations).
* Both images with 0.2 and 0.4 voxel sizes will be reviewed.
* For proper visualization of the mandibular canal, the reference lines will be rotated, so that it lies perpendicular to the mandibular foramen on the axial cuts. Then, scrolling through the corrected sagittal cuts will be performed to review the clearest cut of the full course of the mandibular canal. Moreover, corrected coronal cuts will be reviewed, to determine the exits of the accessory branches (buccal or lingual) if present.
* CBCT images will be interpreted by two oral and maxillofacial radiologists (with different experiences) independently; blinded from demographic data of the patients and from the results of each other.
* The classification of Naitoh et al 2009 will be followed for the categorization of the accessory branches:

  1. Forward canal: emerging from the superior wall of the main canal.
  2. Bucco-lingual canal: emerging from the buccal or the lingual wall of the main canal.
  3. Dental canal: the end of the bifid canal is at the root apex of the molars.
  4. Retromolar canal: emerging from the main canal, opening at the retromolar foramen in the retromolar area.
* Each radiologist will evaluate the images for presence of bifid canal twice with a time lag of two weeks between the two reading sessions. If present, its configuration (classification) will be registered. Any disagreement will be solved by consensus between the two observers.
* If adherence or closeness of the canals to the teeth is detected, then the distance between the canal and the involved tooth will be measured using built in measuring tool in the software.
* The measurements will be carried out by one observer (EE) and will be repeated 2 weeks later for intra-observer reliability assessment.

Bias

No source of bias.

Study Size:

The aim of the study is to assess the prevalence of bifid mandibular canal in Egyptian population. Based on the previous paper by Afsa and Rahmati 2017, the prevalence of bifid mandibular canal was 31% Using a precision of 5, a design effect set at 1 with 95% CI (confidence interval), a total sample size of 329 hemimandibles will be sufficient. The sample size was calculated by Epi info 7 software.

Quantitative Variables:

Quantitative data: The distance between the canal and involved teeth and will be reported as mean and standard deviation.

Statistical methods:

Data will be analyzed using SPSS® v. 15 (SPSS Inc., Chicago, IL) software program. Pearson Chi square and t-tests was performed for statistical analysis among gender, localization and measurements. Categorical data will be described as numbers and percentages. A p value of <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Age range from 18 to 70
* Scans showing the premolar, molar, retromolar areas.

Exclusion Criteria:

* Patients with mandibular lesions.
* Scans with severe metallic artifacts.
* Patients with previous fractures or surgeries.
* Severe bone resorption.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Egyptian population
Sampling Method: Probability Sample
Enrollment: 329 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Bifid mandibular canal detection, measuring device is CBCT software Romexis, measuring unit is percentage ( Dichotomous data - Yes or No ) | up to 2019
  Detection of bifid mandibular canal in Egyptian population

SECONDARY OUTCOMES:
Prevalence of types,measuring device is CBCT software Romexis, measuring unit is Categorical nominal data(%) | up to 2019
  They are either Forward canal, Bucco-lingual canal , Retromolar canal, Dental canal

OTHER OUTCOMES:
Distance to adjacent teeth, measuring device is Built-in measuring tool (ruler), measuring unit is mm | up to 2019
  distance to adjacent teeth will be measured
Region of exit of retromolar canal,measuring device is CBCT software Romexis, measuring unit is Categorical nominal data (%) | up to 2019
  They are either buccal or lingual or non-visible
Prevalence according to gender,measuring unit is categorical nominal data (%) | up to 2019
  They are either male or female

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry, Cairo University, Cairo, Egypt